CLINICAL TRIAL: NCT00839748
Title: The Ohio State University Asthma Registry
Status: Withdrawn | Type: Observational
Why Stopped: personnel redeployment
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jonathan Parsons, Professor of Clinical Internal Medicine, Ohio State University
Other Study IDs: 2003H0221
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: asthma; registry for future asthmatic studies; questionnaires; lung function tests
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- asthmatics: asthmatics registry for those interested in future asthma studies

SUMMARY:
The purpose of this study is to collect information in order to identify people who have asthma and who may be good candidates to participate in one of the future asthma studies to be conducted at The Ohio State University Asthma Clinical Research Center.

DETAILED DESCRIPTION:
Patients from The Ohio State University Division of Pulmonary and Critical Care Medicine will be sent a letter explaining the registry and asking about their interest in participating in this registry. The registry and all procedures related to their inclusion will be explained, opportunity to ask questions will be given and a consent document signed prior to any registry activity. Information about the registry will be shared with the community by newspaper ads, Internet postings, word of mouth, flyers, and other pulmonologists in central Ohio. Those potential registrants may choose to make an appointment to complete lung function tests at the Asthma Clinical Research Center.

The registry and all procedures related to their inclusion will be explained, opportunity to ask questions will be given and a consent document signed prior to any registry activity.

Each participant will be asked to provide appropriate (general medical history, asthma history, current medications, past asthma medications, demographic information, weight height, smoking history, allergies, and prior surgeries. Participants will be asked to complete an Asthma Control Questionnaire, which will be scored to determine how well their asthma is controlled. All consented registrants will be given the opportunity to visit The Ohio State University Asthma Clinical Research Center where an extensive lung function test (spirometry) will be provided. At the Asthma Clinical Research Center each registrant will perform at least three lung function efforts, then given two puffs of albuterol (a fast acting medication that opens airways). After a standard waiting period that meets the standards of the American Thoracic Society, a second set of lung function test will be done. The results of the second set of tests will reflect any reversibility in lung function levels, and will serve as an indicator that treatment may improve lung function. All participants will be given copies of all lung function tests, and the results of the test will be explained to them. All study procedures are provided without cost to the registrant.

ELIGIBILITY:
Inclusion Criteria:

* asthma
* must be able to provide medical history

Exclusion Criteria:

* unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
an asthmatic agrees to have their name and information put in the registry will help study staff determine the most likely candidates for each study | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Parsons, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States